CLINICAL TRIAL: NCT01048073
Title: Non-influenza Etiologies of Acute Respiratory Illness in Southeast Asia
Status: Completed | Type: Observational
Sponsor: South East Asia Infectious Disease Clinical Research Network (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); University of Oxford (Other)
Responsible Party: Dr. Pilaipan Puthavathana, PhD / Principal Investigator, Siriraj Hospital Bangkok, Thailand
Other Study IDs: SEA 019
Record Dates: First submitted 2010-01-12; First posted 2010-01-13 (Estimated); Last update posted 2011-05-27 (Estimated); Status verified 2011-05

CONDITIONS: Lower Respiratory Tract Infection
Keywords: lower respiratory tract infection; non influenza; PCR assay

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * nose swab
  * throat swab
  * nasopharyngeal aspirate
  * nasal wash
  * tracheal aspirate
  * bronchoalveolar lavage
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Acute respiratory infection (ARI) constitutes a leading cause of morbidity, hospitalization and mortality worldwide. The most common etiologic agents of ARI's, especially in children, are viruses.

The study objective is to determine the viral and bacterial etiologies of ARIs in patients with lower respiratory tract infection in South East Asia.

This is a laboratory based surveillance study, in which the archival specimens from hospitalized patients will be tested for respiratory pathogens other than influenza viruses Standard descriptive statistics will be used to present the findings

DETAILED DESCRIPTION:
This study will test 1400 specimens from 1200 patients at the following laboratories:

* National Hospital of Pediatrics, Hanoi
* National Institute of Infectious and Tropical Diseases, Hanoi
* Siriraj Hospital, Bangkok
* National Institute of Health Research and Development, Jakarta
* Hospital for Tropical Diseases, HCMC
* Children Hospital #1, Ho Chi Minh City
* Children Hospital #2, Ho Chi Minh City
* Queen Sirikit National Institute of Child Health

ELIGIBILITY:
Inclusion Criteria:

* Adequately stored respiratory specimens obtained from hospitalized patients suspected of lower respiratory tract infection and were tested for influenza.

Exclusion Criteria:

* Specimens stored at insufficient temperature
* Specimen volume is insufficient
* No demographic data available
* Specimen unsuitable for testing for other technical reasons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with lower respiratory tract infection and were tested for influenza. These patients are admitted to South East Asia Influenza Clinical Research Network hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2010-05; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
the viral and bacterial etiologies of ARIs in patients with lower respiratory tract infection | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pilaipan Pilaipan Puthavathana, MD, Ph.D, Principal Investigator — Siriraj Hospital, Bangkok, Thailand
Locations (9):
- National Institute of Health Research and Development, Jakarta, Indonesia
- Thailand (2):
  - Queen Sirikit National Institute of Child Health, Bangkok
  - Siriraj Hospital, Bangkok
- Vietnam (6):
  - National Hospital of Pediatrics, Hanoi
  - National Hospital of Tropical Diseases, Hanoi
  - Oxford University Clinical Research Unit, Hanoi
  - Children's Hospital No 1, Ho Chi Minh City
  - Children's Hospital No 2, Ho Chi Minh City
  - Hospital for Tropical Diseases, Ho Chi Minh City

REFERENCES:
- [Background] I P M, Nelson EA, Cheuk ES, Leung E, Sung R, Chan PK. Pediatric hospitalization of acute respiratory tract infections with Human Bocavirus in Hong Kong. J Clin Virol. 2008 May;42(1):72-4. doi: 10.1016/j.jcv.2007.12.016. Epub 2008 Mar 4. PMID 18296108
- [Background] Tsang KW, File TM Jr. Respiratory infections unique to Asia. Respirology. 2008 Nov;13(7):937-49. doi: 10.1111/j.1440-1843.2008.01409.x. PMID 18945321
- [Background] Yuan XH, Jin Y, Xie ZP, Gao HC, Xu ZQ, Zheng LS, Zhang RF, Song JR, Hou YD, Duan ZJ. Prevalence of human KI and WU polyomaviruses in children with acute respiratory tract infection in China. J Clin Microbiol. 2008 Oct;46(10):3522-5. doi: 10.1128/JCM.01301-08. Epub 2008 Jul 30. PMID 18667596
- [Background] Drews SJ, Blair J, Lombos E, DeLima C, Burton L, Mazzulli T, Low DE. Use of the Seeplex RV Detection kit for surveillance of respiratory viral outbreaks in Toronto, Ontario, Canada. Ann Clin Lab Sci. 2008 Autumn;38(4):376-9. PMID 18988931
- [Background] Roh KH, Kim J, Nam MH, Yoon S, Lee CK, Lee K, Yoo Y, Kim MJ, Cho Y. Comparison of the Seeplex reverse transcription PCR assay with the R-mix viral culture and immunofluorescence techniques for detection of eight respiratory viruses. Ann Clin Lab Sci. 2008 Winter;38(1):41-6. PMID 18316781
- [Background] Yoo SJ, Kuak EY, Shin BM. Detection of 12 respiratory viruses with two-set multiplex reverse transcriptase-PCR assay using a dual priming oligonucleotide system. Korean J Lab Med. 2007 Dec;27(6):420-7. doi: 10.3343/kjlm.2007.27.6.420. PMID 18160832